CLINICAL TRIAL: NCT02788136
Title: Analisi Del Profilo Sierico Steroideo Basale e Dopo Stimolo Con Gonadotropina Corionica Umana (HCG) Nei Soggetti Affetti da Sindrome di Klinefelter (SK).
Brief Title: Human Chorionic Gonadotropin Stimulation Effects on Steroidogenesis in Men With Klinefelter Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda USL Modena (Other)
Responsible Party: Principal Investigator, Manuela Simoni, Ordinary Professor, Azienda USL Modena
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: Klinefelter & hCG
Record Dates: First submitted 2016-05-30; First posted 2016-06-02 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2016-06

CONDITIONS: Steroidogenesis; Klinefelter Syndrome; Human Chorionic Gonadotropin (hCG) Stimulation
MeSH Terms: conditions — Klinefelter Syndrome | interventions — Chorionic Gonadotropin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Klinefelter syndrome (Experimental): 13 men with diagnosis of Klinefelter syndrome were stimulated with human chorionic gonadotropin (hCG)
  Interventions: Drug: human chorionic gonadotropin
- Control (Active Comparator): 12 healthy age-related men were stimulated with human chorionic gonadotropin (hCG)
  Interventions: Drug: human chorionic gonadotropin

INTERVENTIONS:
Drug: human chorionic gonadotropin — At 08 AM of day 0, all subjects underwent to a single intramuscular injection of hCG of 5000 IU
  Other Names: hCG

SUMMARY:
The study design included six visits. During the first visit (visit 0), the subjects underwent physical examination(height, weight, body mass index (BMI), arm span, and upper segment measurement) and testicular ultrasound (US) for the calculation of testicular volume. At 0800 h of day 0, all subjects provided a basal blood sample immediately followed by a single intramuscular injection of hCG of 5000 IU. Further five visits were performed each of five following consecutive days after the hCG injection. A blood sample was taken at each visit after an overnight fast

DETAILED DESCRIPTION:
Blood samples were centrifuged at 2955 g for 15 min. Sera were transferred into plain polypropylene tubes and stored at -20°C until assayed. P, 17OHP, AS, DHEA, and TS were determined by LC-MS/MS at the laboratory of the Centre for Applied Biomedical Research of the S. Orsola-Malpighi Hospital, Alma Mater Studiorum, University of Bologna, Bologna, Italy.

ELIGIBILITY:
Inclusion Criteria:

* Klinefelter syndrome diagnosis at kariotype evaluation for the study group
* Healthy age-matched men in the control group

Exclusion Criteria:

* previous or ongoing androgen therapy

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2012-02; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Testosterone | visit 1 (Day 1)
  Using mass spectrometry

SECONDARY OUTCOMES:
Testicular volume | visit 0 (Baseline)
  testicular volume at ultrasonography
Steroids | Visit 0 (Baseline)
  Steroidogenesis evaluated through mass spectrometry
Steroids | Visit 1 (Day 1)
  Steroidogenesis evaluated through mass spectrometry
Steroids | Visit 2 (Day 2)
  Steroidogenesis evaluated through mass spectrometry
Steroids | Visit 3 (Day 3)
  Steroidogenesis evaluated through mass spectrometry
Steroids | Visit 4 (Day 4)
  Steroidogenesis evaluated through mass spectrometry
Steroids | Visit 5 (Day 5)
  Steroidogenesis evaluated through mass spectrometry

CONTACTS AND LOCATIONS:
Locations (1):
- AziendaUSLModena, Modena, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Belli S, Santi D, Leoni E, Dall'Olio E, Fanelli F, Mezzullo M, Pelusi C, Roli L, Tagliavini S, Trenti T, Granata AR, Pagotto U, Pasquali R, Rochira V, Carani C, Simoni M. Human chorionic gonadotropin stimulation gives evidence of differences in testicular steroidogenesis in Klinefelter syndrome, as assessed by liquid chromatography-tandem mass spectrometry. Eur J Endocrinol. 2016 Jun;174(6):801-11. doi: 10.1530/EJE-15-1224. PMID 27188454